CLINICAL TRIAL: NCT01638585
Title: Patients With Diabetic Foot Syndrome and Critical Limb Ischemia - a Randomized Clinical Trial With Urokinase
Brief Title: Safety and Efficacy Study of Urokinase for the Treatment of Diabetic Foot Syndrome and Critical Limb Ischemia
Acronym: August2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruition number was not reached
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: August 2; 2010-023426-20 (EudraCT Number)
Record Dates: First submitted 2012-05-14; First posted 2012-07-11 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Foot; Critical Limb Ischemia
MeSH Terms: conditions — Diabetic Foot; Chronic Limb-Threatening Ischemia | interventions — Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard therapy (No Intervention): patients receiving standard therapy for diabetic foot syndrome with critical limb ischemia, i. e. structured therapy of lesions with antibiosis, pressure relief and therapy of risk factors according to the relevant guidelines.
- urokinase (Active Comparator): patients receiving urokinase short infusions in addition to standard therapy
  Interventions: Drug: urokinase

INTERVENTIONS:
Drug: urokinase — daily short infusions, i. e. i. v. application of 1.000.000 I.E. urokinase over 30 min. for at least 10 and up to 21 days during the 30 days after randomization
  Other Names: Urokinase HS medac
  Arms: urokinase

SUMMARY:
In this randomized clinical trial (RCT) the investigators are trying to find out whether a low-dose therapy with daily short infusions of urokinase using 10 to 21 doses over a maximum of 30 days is capable of prolonging the survival time without major amputation.

DETAILED DESCRIPTION:
August-2 is a trial embedded in the August-1 registry study. All patients enrolled in August-2 are also part of August-1, but there will be patients who are documented in the register, but will not take part in August-2. The investigators want to find out to which extent the patients in the registry are representative to the overall population suffering from this condition and how the therapeutic success of other therapy regimes can be described.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* angiopathic or angioneuropathic critical limb ischemia (at least Wagner-Armstrong stadium II)
* participation in the August-1 Register
* revascularization not possible or residual ischemia after revascularization
* persisting ulcerations despite antibiosis, adjustment of blood glucose levels and debridement
* expected further hospitalization for at least 3 weeks (pressure relief and antibiosis)
* fibrinogen >= 4g/l
* signed informed consent

Exclusion Criteria:

* life expectancy < 1 year
* prior major amputation
* planned major amputation
* prior therapy of the current episode of diabetic foot syndrome with urokinase (except in cases of revascularization when the duration between the intervention and randomization must not exceed 7 days)
* mechanical heart valve substitute
* cerebral event with CT-detectable changes in the last 3 months
* non-remediated proliferation retinopathy
* uncontrolled hypertension (systolic >180 mmg, diastolic >100 mmHg)
* hemorrhagic diathesis (spontaneous quick < 50%, spontaneous PTT > 40 s, thrombocytes < 100 Gpt/l)
* gastrointestinal bleeding or ulcers in the last 4 weeks
* prior reverse bypass operation
* contraindications against therapy with urokinase acc. to the SMPc
* concurrent participation in another clinical trial
* insufficient compliance
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Duration of survival without major amputation in urokinase group compared to group with standard therapy | within the FU of 12 months

SECONDARY OUTCOMES:
total mortality | 12 months after randomization
minor amputation | 12 months after randomization
Number of necessary revisions in case of minor amputation | 12 months after randomization
complete healing of targeted lesion | within the FU of 12 months
new lesions on previously affected leg | within the FU of 12 months
efficacy in dialysis patients | within the FU of 12 months
duration of hospital stay | from baseline examination until first release (expected average of 2 weeks in general)
re-hospitalization after dismissal following end of therapy with urokinase | within the FU of 12 months
Necessity for parenteral therapy with vasoactive substances | from baseline to end of 12 months FU
  During the follow-up it will be documented wether the administration of parenterally applied vasoactive substances or thrombocyte aggregation inhibitors was necessary.
cardiovascular events | from baseline to end of 12 months FU
  Any major cardiovascular events during the follow-up period. Duration, severity, outcome and causal relationship with urokinase therapy will be documented.
incidence and type of bleeding events | from randomization until day 33
incidence and type of other adverse events | from baseline to end of 12 months FU
new lesions on the contralateral leg | within the FU of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: S. Schellong, Prof.Dr.med., Principal Investigator — Städt. KH Dresden-Friedrichstadt
Locations (18):
- Germany (18):
  - Diabetes Klinik, Bad Mergentheim
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Ev. KH Königin Elisabeth Herzberge, Berlin
  - Martin-Luther-Krankenhaus, Berlin
  - Klinikum Bielefeld gGmbH, Bielefeld
  - Stiftungsklinikum Mittelrhein, Boppard
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Dortmund gGmbH, Dortmund
  - Städtisches Krankenhaus DD-Neustadt, Dresden
  - Krankenhaus Dresden-Friedrichstadt, Dresden
  - Uniklinikum "Carl Gustav Carus" der TU Dresden, Dresden
  - Weißeritztal Kliniken GmbH, Freital
  - Asklepios Westklinikum, Hamburg
  - Universitätsklinikum Leipzig AöR, Leipzig
  - HELIOS Krankenhaus, Leisnig
  - Klinikum Westfalen/Klinikum am Park, Lünen
  - Klinikum Stuttgart, Bürgerhospital, Stuttgart
  - KH der Barmherzigen Brüder, Trier